CLINICAL TRIAL: NCT06463795
Title: Effects of Transcranial Direct Current Stimulation on Lower Limb Performance in Stroke Patients
Brief Title: tDCS and Lower Limb Performance in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC01898 Saira Muzaffar Shah
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Stroke; Lower limb; transcranial direct current stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS Group (Experimental): Electrode placement: Anodal electrode placed over primary motor cortex area (M1) while the cathode placed over contralateral orbit.
  Duration of 20 minutes with intensity of 2mA, ramping up and down at 8 seconds. the density of 0.07 C/cm2 for 3 days/week for 8 weeks
  Interventions: Device: tDCS
- Sham Group (Sham Comparator): Electrode placement: Anodal electrode placed over primary motor cortex area (M1) while the cathode placed over contralateral orbit.
  Duration of 20 minutes with intensity of 0.5mA, ramping up and down at 150 and 30 seconds respectively. There will be brief stimulation period of 3-5% active session duration the density of 0.07 C/cm2 for 3 days/week for 8 weeks
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: tDCS — active anodal tDCS
  Arms: tDCS Group
Device: Sham tDCS — sham anodal tDCS
  Arms: Sham Group

SUMMARY:
Lower limb rehabilitation is especially important, as the simple act of regaining the ability to walk has subsequent effects on the ability to engage in activities of daily living .So, this study will contribute in describing the management of lower limb motor recovery along with the therapeutic intervention (MRP) with tDCS (anodal stimulation). This study aims to address some of the drawbacks observed in previous studies like allocation concealment, small sample size due to drop outs, short term effects of tDCS and experimental designs as well.

DETAILED DESCRIPTION:
Transcranial Direct Current Stimulation (tDCS) appears to be an intriguing adjuvant for stroke neurorehabilitation, though there are many other methods available. Depending on the polarity used, tDCS alters cortical excitability when electrodes applied over the motor cortex area (M1) to be stimulated, and the cathode above the contralateral eye (Orbital area), tDCS (thus termed anodal) increases cortical excitability. It is easy to use, safe and has minimal side effects like a sensation of itching, post-stimulation headache and sometimes mild nausea may experience. Numerous research indicates that cortical activity rises in conjunction with gait. According to a number of studies, corticospinal neuron activity either parallels or possibly even partially regulates the activity of spinal motor neurons during walking. There exist various techniques for implementing transcranial direct current stimulation in conjunction with multiple supplementary therapies.

ELIGIBILITY:
Inclusion Criteria:

* Stroke for more than 6 months.
* National Institutes of Health Stroke Scale (NIHSS) for severity level (Mild (1-4), Moderate (5-15), Moderate to Severe (16-20), Severe (21-42)

Exclusion Criteria:

* Epilepsy
* Scalp injury/ skin lesion e.g. psoriasis or eczema etc.
* Patient with lower limb amputation or any MSK/neurological disorder that limit the LE function
* Implanted medical devices including intracranial electrodes, surgical clips, shrapnel or a pacemaker

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
FMA-lower extremity | 8 week
  FMA-LE is a method used to measure motor function, balance, and function of joints in post-stroke patients. Fugl Meyer Assessment of Lower Extremity (FMA-LE). FMA-LE is a method used to evaluate the performance of motor movement on the lower limbs (hips, knees, feet, and ankles) and predicts recovery function of motion in stroke patients. FMA-LE method consists of 17 items are organized into several sub-sections, namely reflection part, synergistic part, and coordination with Mild (˃45),Moderate (30-45),Severe (˂30) scores(12). It shows sensitivity of 0.87 and specificity of 0.81
Six Minute walk Test | 8 week
  The Six-Minute Walk Test (6MWT) is a functional walking test in which the distance that a stroke patient can walk within six minutes is evaluated. This test has been used to assess individuals with stroke, head injury and Parkinson's disease. There are no actual items to the 6MWT.It is a simple test that requires a 100-ft, quiet, indoor, flat, straight rectangular hallway. The walking course must be 30m in length. The length of the 30m corridor must be marked by colored tape at every 3m. The turnaround must be marked with a cone. Some studies have used 20 and 50m corridors. It has excellent test-retest reliability (0.99 distance in meters) among stroke survivors

SECONDARY OUTCOMES:
Stroke Specific Quality of Life | 8 week
  The Stroke Specific Quality Of Life scale (SS-QOL) is a patient-centered outcome measure intended to provide an assessment of health-related quality of life specific to patients with stroke. It is a self-report scale containing 49 items in 12 domains including Energy, Mobility, Upper extremity function, Work/productivity, Mood, Self-care, Social roles, Family roles, Vision, Language, Thinking, and Personality. Score ranges from 49 to 245. Higher scores indicate better QOL(14).It has a sensitivity of 70.0% and a specificity of 75.8%

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411
- [Background] Clark B, Whitall J, Kwakkel G, Mehrholz J, Ewings S, Burridge J. The effect of time spent in rehabilitation on activity limitation and impairment after stroke. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD012612. doi: 10.1002/14651858.CD012612.pub2. PMID 34695300
- [Background] Bai X, Guo Z, He L, Ren L, McClure MA, Mu Q. Different Therapeutic Effects of Transcranial Direct Current Stimulation on Upper and Lower Limb Recovery of Stroke Patients with Motor Dysfunction: A Meta-Analysis. Neural Plast. 2019 Nov 16;2019:1372138. doi: 10.1155/2019/1372138. eCollection 2019. PMID 31827495